CLINICAL TRIAL: NCT02105454
Title: A Phase II Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 + MK-8742 + Ribavirin (R) in Subjects With Chronic Hepatitis C Virus Infection Who Failed Prior Direct Acting Antiviral Therapy
Brief Title: Study of Grazoprevir (MK-5172) + Elbasvir (MK-8742) + Ribavirin in Participants With Chronic Hepatitis C Who Failed Prior Direct-Acting Antiviral Therapy (MK-5172-048)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5172-048; 2013-004213-41 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GZR 100 mg + EBR 50 mg + RBV for 12 weeks (Experimental): Participants receive grazoprevir 100 mg once per day (QD), elbasvir 50 mg QD, and RBV 800 - 1400 mg total daily dose divided twice per day (based on body weight) for 12 weeks
  Interventions: Drug: Grazoprevir (GZR); Drug: Elbasvir (EBR); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Grazoprevir (GZR) — 100 mg oral tablet (total daily dose)
Drug: Elbasvir (EBR) — 10 mg oral capsule (total daily dose = 5 capsules)
Drug: Ribavirin (RBV) — 200 mg oral capsule (total daily dose = 4-7 capsules)

SUMMARY:
In this study, participants with hepatitis C virus (HCV) genotype 1 (GT1) who failed prior direct-acting antiviral (DAA) therapy will receive Grazoprevir (MK-5172) + Elbasvir (MK-8742) + Ribavirin (RBV) to evaluate sustained virologic response (SVR) using this drug combination.

ELIGIBILITY:
Inclusion criteria:

* Documented chronic HCV GT1 infection (with no evidence of non-typable or mixed genotype)
* Absence of cirrhosis, or cirrhosis with these criteria: METAVIR F4, or Fibroscan with result >12.5 kPa, or FibroSure® (Fibrotest®) score of >0.75 + aspartate aminotransferase (AST): platelet ratio index (APRI) of >2- Prior regimen containing an approved DAA (boceprevir, telaprevir, simeprevir, or sofosbuvir), pegylated interferon, and/or RBV
* Participants of reproductive potential must agree to remain truly abstinent or use (or have their partner use) 2 acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations

Exclusion criteria:

* Received any HCV regimen containing a DAA with the exception of boceprevir, telaprevir, simeprevir, or sofosbuvir in combination with pegylated interferon and/or RBV
* Evidence of decompensated liver disease or cirrhosis
* Co-infected with hepatitis B virus or human immunodeficiency virus (HIV)
* History of malignancy <=5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or under evaluation for other active or suspected malignancy
* Evidence of hepatocellular carcinoma (HCC) or under evaluation for HCC
* Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study
* Clinically-relevant drug or alcohol abuse within 12 months of screening
* Pregnant, breast-feeding, or expecting to conceive or donate eggs or sperm from at least 2 weeks prior to Day 1 and continue throughout treatment and follow up, or longer if dictated by local regulations
* Male participant whose female partner (s) is/are pregnant
* Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* Poor venous access
* History of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorders (e.g., celiac sprue disease)
* Hemoglobinopathy, including, but not limited to, thalassemia major
* Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* Evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Forns X, Gordon SC, Zuckerman E, Lawitz E, Calleja JL, Hofer H, Gilbert C, Palcza J, Howe AY, DiNubile MJ, Robertson MN, Wahl J, Barr E, Buti M. Grazoprevir and elbasvir plus ribavirin for chronic HCV genotype-1 infection after failure of combination therapy containing a direct-acting antiviral agent. J Hepatol. 2015 Sep;63(3):564-72. doi: 10.1016/j.jhep.2015.04.009. Epub 2015 Apr 18. PMID 25895428
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518
- [Derived] Buti M, Gordon SC, Zuckerman E, Lawitz E, Calleja JL, Hofer H, Gilbert C, Palcza J, Howe AY, DiNubile MJ, Robertson MN, Wahl J, Barr E, Forns X. Grazoprevir, Elbasvir, and Ribavirin for Chronic Hepatitis C Virus Genotype 1 Infection After Failure of Pegylated Interferon and Ribavirin With an Earlier-Generation Protease Inhibitor: Final 24-Week Results From C-SALVAGE. Clin Infect Dis. 2016 Jan 1;62(1):32-6. doi: 10.1093/cid/civ722. Epub 2015 Sep 14. PMID 26371152

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following 12 weeks of treatment with grazoprevir (GZR), elbasvir (EBR) and ribavirin (RBV), participants were followed-up for an additional 24 weeks.
Period: Overall Study
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Started | 79
Completed | 78
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response (SVR) at 12 Weeks After the End of All Study Therapy (SVR12)
Description: SVR12 is defined as participants having hepatitis C virus ribonucleic acid (HCV RNA) level lower than the limit of quantification (LLoQ, <15 IU/mL in plasma), either target detected and unquantifiable or undetectable 12 weeks after the end of all study therapy.
Time Frame: Up to 24 weeks
Population: Per protocol population excludes participants due to important deviations from the protocol that may substantially affect the results of the primary and key secondary efficacy endpoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Number analyzed (Participants) | 70
Percentage of participants | 97.1 [90.1 to 99.7]

2. Primary Outcome: Percentage of Participants Experiencing Adverse Events
Description: Adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product.
Time Frame: Up to 40 weeks (from Day 1 [post-dose] through 24 [-12/+4] weeks following last dose of study drug)
Population: All participants as treated population defined as all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Number analyzed (Participants) | 79
Percentage of participants | 79.7 [69.2 to 88.0]

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 12 weeks
Population: All participants as treated population defined as all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Number analyzed (Participants) | 79
Percentage of participants | 1.3 [0.0 to 6.9]

4. Secondary Outcome: Percentage of Participants Achieving SVR12 by Prior Direct-acting Antiviral (DAA) Therapy
Description: SVR12 is defined as participants having HCV RNA level lower than the LLoQ (<15 IU/mL in plasma), either target detected and unquantifiable or undetectable 12 weeks after the end of all study therapy. Prior DAA therapy regimen included boceprevir, telaprevir, simeprevir, or sofosbuvir taken concomitantly with peginterferon and ribavirin. Below categories specify with our without resistance-associated variants (RAVs) of the hepatitis C virus.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Number analyzed (Participants) | 70
Percentage of participants
  Boceprevir with signature baseline RAVs, n=9 | 88.9 [51.8 to 99.7]
  Boceprevir without signature baseline RAVs, n=16 | 100.0 [79.4 to 100.0]
  Telaprevir with signature baseline RAVs, n=18 | 94.4 [72.7 to 99.9]
  Telaprevir without signature baseline RAVs, n=22 | 100.0 [84.6 to 100.0]
  Simeprevir with signature baseline RAVs, n=4 | 100.0 [39.8 to 100.0]
  Simeprevir without signature baseline RAVs, n=1 | 100.0 [2.5 to 100.0]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): up to 40 weeks (including 24-week follow-up [-12/+4 weeks]); non-serious adverse events (NSAEs): Up to 14 weeks (including 2-week follow-up)
Description: All participants as treated population included all participants who received at least 1 dose of study medication. MedDRA version 17.1: AEs summarized in the 1st Clinical Study Report (CSR) (through at least 12 weeks of follow-up); MedDRA version 18.0: AEs summarized in the final CSR after study completion (through 24 weeks of follow-up).
Arm/Group | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 6/79
Other Adverse Events (participants affected / at risk) | 47/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks (N=79)
Appendicitis (Infections and infestations) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GZR 100 mg + EBR 50 mg + RBV for 12 Weeks (N=79)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (11)
Nausea (Gastrointestinal disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 12 (12)
Fatigue (General disorders) | 22 (24)
Haemoglobin decreased (Investigations) | 4 (4)
Headache (Nervous system disorders) | 15 (16)
Insomnia (Psychiatric disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.